CLINICAL TRIAL: NCT00352742
Title: A Phase I/II Study of ATN-224 and Bortezomib in Patients With Multiple Myeloma Relapsed From or Refractory to Bortezomib
Brief Title: A Study of ATN-224 and Bortezomib in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Attenuon (Industry)
Responsible Party: Jennifer Callahan, Senior Manager, Clinical Development, Attenuon, LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATN-224-007
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; bortezomib; ATN-224; refractory; relapsed; antiangiogenic
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — tetrathiomolybdate; Bortezomib

ARMS (1):
- 1 (Experimental): ATN-224 + bortezomib
  Interventions: Drug: ATN-224 + bortezomib

INTERVENTIONS:
Drug: ATN-224 + bortezomib — ATN-224 and bortezomib dose to be determined in Phase I portion of study

SUMMARY:
The purpose of this study is to describe the safety and effect of ATN-224 in combination with bortezomib (Velcade®) in patients with Multiple Myeloma who are relapsed from or refractory to bortezomib.

DETAILED DESCRIPTION:
Multiple myeloma is a bone marrow based malignancy of plasma cells that is highly treatable but rarely curable. Angiogenesis, defined as the growth of new blood vessels from pre-existing vessels, is a requirement for the growth of nearly all tumors. An increase in bone marrow angiogenesis is present in Multiple Myeloma and correlates with disease progression. Several new therapies that target angiogenic pathways have shown clinical efficacy. ATN-224 is a small molecule that has been shown in pre-clinical studies to be antiangiogenic.

Using one agent to overcome resistance of another agent is a treatment regimen used in oncology. A preclinical study with the combination of ATN-224 and bortezomib shows that the combination is more effective than either single agent in a bortezomib resistant cell line.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed multiple myeloma that has been treated with at least one different prior anti-myeloma regimens including one with bortezomib and is currently showing evidence of progressive disease
2. Myeloma that is refractory to the most recent bortezomib-containing regimen as demonstrated by progressive disease while on bortezomib or that relapsed within 12 weeks of the last dose of bortezomib either as a single agent or in combination with other agents
3. Measurable disease defined as a serum M-protein concentration on electrophoresis ≥1 g/dL of IgG myeloma or ≥0.5 g/dL of IgA myeloma or IgM myeloma or urinary excretion of monoclonal light chain ≥200 mg/24 hours
4. Age >18 years
5. Life expectancy of greater than 3 months
6. ECOG performance status <2 (Karnofsky >60%; see Appendix A)
7. Adequate organ and marrow function as defined below:

   * absolute neutrophil count ≥1,000/uL
   * platelets ≥75,000/uL
   * hemoglobin ≥8 g/dL
   * total bilirubin ≤2 X institutional upper limit of normal (ULN)
   * AST(SGOT) and ALT(SGPT) ≤3 X ULN
   * creatinine clearance ≥30 mL/min (measured or calculated)

   Patients are allowed to receive blood transfusions before receiving their first dose of ATN-224 to bring the hemoglobin level to ≥8 g/dL to meet eligibility criteria.
8. Use of adequate contraception. The effects of ATN 224 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because antiangiogenic agents are known to be teratogenic, women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal and/or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation through the follow up visit 28 days after the last dose of ATN 224.
9. Willingness to forego taking copper- or zinc-containing vitamins or supplements
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or thalidomide, lenalidomide, dexamethasone, arsenic trioxide, bortezomib, or glucocorticosteroids within 3 weeks prior to the first dose of ATN-224 or failure to recover from reversible adverse events due to agents administered previously
2. Patients who cannot tolerate, based on previous experience, the assigned dose of bortezomib, including those with ≥ Grade 2 neuropathy
3. Concurrent administration of any other investigational agents
4. History of malabsorption syndromes or other gastrointestinal disorders that may affect ATN-224 absorption, including bowel obstruction, celiac disease, sprue, cystic fibrosis
5. Ineligible to receive omeprazole (Prilosec® OTC) or other long-acting antacid
6. Inability to swallow study medication capsules
7. Not a suitable candidate in the opinion of the investigator for additional bortezomib therapy
8. Other serious medical or psychiatric illness preventing informed consent or intensive treatment
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
10. Women who are pregnant or lactating
11. Known history of HIV
12. History of another prior cancer, except basal cell carcinoma or carcinoma in situ of the cervix (or if there has been no evidence of recurrence for at least 5 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-09 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Phase I: Determine a safe dose of ATN-224 and bortezomib to be used in the phase II portion of the study | Ongoing
Phase II: Efficacy | End of Study

SECONDARY OUTCOMES:
Phase I: Preliminary evidence of efficacy | End of Study
Phase II: progression-free survival and duration of response | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Gordon, MD, Study Director
Locations (10):
- United States (10):
  - Hematolgy-Oncology Medical Group of Fresno, Inc., Fresno, California
  - Institute for Myeloma and Bone Cancer Research, West Hollywood, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Billings Clinic, Billings, Montana
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - SUNY Downstate, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas